CLINICAL TRIAL: NCT02499939
Title: Ultrasound Therapy and Therapeutic Exercise for Chemotherapy Induced Peripheral Neuropathy (CIPN) in Colon and Colorectal Cancer Patients: A Randomized Controlled Pilot Trial
Brief Title: Ultrasound Therapy and Therapeutic Exercise for Chemotherapy Induced Peripheral Neuropathy (CIPN)
Acronym: ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margie McNeely (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Margie McNeely, Associate Professor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA-CC-15-0107
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-04

CONDITIONS: Colon Neoplasms; Colorectal Neoplasms
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Standard of Care; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Participants in this group will receive standard education about CIPN and therapeutic exercises to carry out at home.
  Interventions: Behavioral: Standard Care
- Experimental: Ultrasound Therapy (Experimental): Participants in this group will receive standard education about CIPN and therapeutic exercises to carry out at home. Participants in this group will also undergo 10 daily treatments of ultrasound therapy (e.g., Monday to Friday for two weeks) that is administered to their toes and fingers. The ultrasound therapy will be administered over the first two weeks of the intervention period.
  Interventions: Behavioral: Standard Care; Other: Ultrasound Therapy

INTERVENTIONS:
Behavioral: Standard Care — Education and home exercises
Other: Ultrasound Therapy — Ultrasound is a therapeutic modality that is used by physical therapists to help reduce local tissue pain and inflammation. Ultrasound is applied using a round-headed wand or probe that is placed in direct contact with the patient's skin. Ultrasound gel is used on all surfaces of the ultrasound head to reduce friction and assist in the transmission of the ultrasonic waves. For the purposes of treatment for CIPN, the ultrasound will be applied for 5 minutes to each limb (right toes, left toes, right fingers, left fingers) at frequency of 3.0 megahertz (MHz) and an intensity of 0.7-0.8 watts per cm2.
  (For CIPN, the ultrasound will be administered at a lower intensity in order to avoid a heating effect on the tissues.)
  Arms: Experimental: Ultrasound Therapy

SUMMARY:
The primary purpose of the trial is to determine the preliminary efficacy of therapeutic ultrasound in the treatment of pain and sensory disturbance related to chemotherapy induced peripheral neuropathy.

DETAILED DESCRIPTION:
Thirty cancer patients with colon or colorectal cancer undergoing chemotherapy treatment including the agent oxaliplatin will take part in the study. Patients will be randomly assigned to either standard care alone (education and therapeutic exercises) or standard care plus 10 treatments of therapeutic ultrasound to the toes and fingers.

Participants in both groups will follow a home exercise program for a 6 week period. Therapeutic ultrasound will be administered daily (e.g., Monday to Friday) over the first two week period of the study.

ELIGIBILITY:
Inclusion Criteria:

1. adults18 or older,
2. receiving or have received chemotherapy treatment for colon or colorectal cancer,
3. chemotherapy regimen includes the agent oxaliplatin,
4. Grade 1, 2 or 3 on the National Cancer Institute Common Terminology Criteria for Adverse Events for sensory and motor neuropathy.

Exclusion Criteria:

1. neuropathy pre-existing the patient's cancer diagnosis;
2. contraindications to therapeutic ultrasound:

   * active cancer in region of hands or feet,
   * presence of deep vein thrombosis,
   * lack of sensation in hands or feet,
   * metal or plastic implants in hands or feet;
3. peripheral vascular disease or other serious existing non-malignant disease which may affect their ability to complete testing and treatment sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy Gynecological Oncology Group Neurotoxicity-12 item scale | 6 weeks
  Change in pain and sensory disturbance

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-CIPN twenty-item scale (QLQ-CIPN20)3 | 6 weeks
  Change in quality of life and symptoms related to chemotherapy induced peripheral nerve injury
Protective sensation | 6 weeks
  Change in protective sensation: using a 10g monofilament for the feet and 6g for the hands to determine presence or absence of protective sensation.
Temperature sensation | 6 weeks
  Change in temperature sensation: hot and cold test tubes will be applied to the feet and hands to determine ability to distinguish hot and cold sensations.
Vibration sensation | 6 weeks
  Change in vibration sensation: A 128 Hz tuning fork will be applied to the big toe, medial malleolus, thumb and ulnar styloid to determine presence/ absence of vibration sensation.
Reflexes | 6 weeks
  Change in reflexes: The reflex of the Achilles tendon will be tested to determine the presence/ absence of this tendon reflex
Balance Assessment | 6 weeks
  Change in two foot and single foot balance: balance will be assessed in two conditions: eyes open and eyes closed.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Yurick, BSc, Principal Investigator — Alberta Health services
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Onazi MM, Yurick JL, Harris C, Nishimura K, Suderman K, Pituskin E, Chua N, McNeely ML. Therapeutic Ultrasound for Chemotherapy-Related Pain and Sensory Disturbance in the Hands and Feet in Patients With Colorectal Cancer: A Pilot Randomized Controlled Trial. J Pain Symptom Manage. 2021 Jun;61(6):1127-1138. doi: 10.1016/j.jpainsymman.2020.10.028. Epub 2020 Nov 1. PMID 33137422